CLINICAL TRIAL: NCT03973736
Title: Impatto Della Revisione Radiologica Con Valutazione Multidisciplinare Nella Gestione Terapeutica Dei Pazienti Affetti da Adenocarcinoma Pancreatico (PAC)
Brief Title: Impact of Multidisciplinary and Radiologic Review on Outcome of Pancreatic Cancer Patients: an Observational Study
Acronym: RevRadPAC
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 286/2018/OSS/AUSLRE
Record Dates: First submitted 2019-05-27; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PDAC patients diagnosed in 2008-2011
- PDAC patients diagnosed in 2013-2016
  Interventions: Other: application of a diagnostic and therapeutic protocol (multidisciplinary discussion and radiological CT review)

INTERVENTIONS:
Other: application of a diagnostic and therapeutic protocol (multidisciplinary discussion and radiological CT review) — Since the introduction of the new protocol in 2012, a single central multidisciplinary team has been formalized, with weekly discussion of cases, including different specialists from all the provincial hospitals. CT scans of discussed cases are reviewed by one of two experienced radiologists based on pre-defined criteria.
  Groups: PDAC patients diagnosed in 2013-2016

SUMMARY:
The investigators compared two different time periods respectively before and after the application of a dedicated diagnostic and therapeutic protocol for pancreatic ductal adenocarcinoma including multidisciplinary discussion and radiological review of cases, in order to evaluate the impact of the new protocol on surgical failures and overall survival.

DETAILED DESCRIPTION:
Since 2012 in Reggio Emilia a new diagnostic and therapeutic protocol has been implemented including multidisciplinary team discussion of non-metastatic PDACs and radiological review of CT scans by an experienced radiologist.

The aim of this study is to measure the impact of this new protocol on the occurrence of surgical failures, including incomplete resection or surgery in which resection resulted impossible at all. The investigators also describe the changes in overall survival and process indicators such as the proportion of patients referred to different therapeutic options (upfront surgery, neoadjuvant chemotherapy and no surgery) and the compliance with referral.

Through a population-based cohort study, the investigators evaluated the impact of the new protocol on therapeutic management and surgical outcome of patients with non-metastatic PDAC by comparing two four-years periods, respectively 2008-2011 and 2013-2016, before and after the introduction of the protocol. Since 2012 was the transitional year when the protocol was introduced, patients diagnosed with PDAC in 2012 were excluded.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive inhabitants of the Reggio Emilia province with incident PDACs in 2008-2011 and 2013-2016 periods

Exclusion Criteria:

* pancreatic cancers with cytohistological diagnosis different from PDAC,
* diagnosis in 2012,
* metastatic disease at diagnosis (stage IV) or unknown stage at diagnosis,
* patients aged >85 years.

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Reggio Emilia Pancreatic Cancer Register registered 1157 PDAC cases from 2008 to 2016. After exclusion of cases diagnosed in 2012, patients aged >85 years and cancer staged as IV or with unknown stage, a total of 132 and 184 patients were included in analysis respectively for 2008-2011 and 2013-2016 periods.
Sampling Method: Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Proportion of surgical failures on the total of eligible patients | immediately after surgery
  proportion of patients with incomplete resection or who received surgery in which resection was not possible

SECONDARY OUTCOMES:
Overall survival | 24 months
  overall survival (restricted to patients with at least 24 months follow-up)
proportion of patients referred to different therapeutic options | up to 1 year
  proportion of patients referred to different therapeutic options (upfront surgery, neoadjuvant chemotherapy and no surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL - IRCCS di Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No